CLINICAL TRIAL: NCT03615651
Title: Probiotic Effects on the Microbe-brain-gut Interaction and Brain Activity During Stress Tasks in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Robert Brummer, Professor, MD, Örebro University, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017/398
Record Dates: First submitted 2018-06-08; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Probiotics; Gut Microbiota; Emotional Stress; Magnetic Resonance Imaging
MeSH Terms: conditions — Stress, Psychological | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): All study participants will receive the study product and the placebo in a randomized, double-blind crossover fashion. Probiotic and placebo products have similar appearance and taste.
  Interventions: Other: Placebo
- Probiotic (Experimental): All study participants will receive the study product and the placebo in a randomized, double-blind crossover fashion. Probiotic and placebo products have similar appearance and taste.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — The Probiotic Formula is commercially available and contains a combination of 3 probiotic strains in addition to other nutrients. The total daily amount of probiotic strain in the product will be no less than 3 billion colony-forming units (CFU) per 3 g powder sachet.
  Arms: Probiotic
Other: Placebo — Placebo intervention.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine if and how the "Probiotic Product" affects functional brain responses in healthy subjects during an emotional- and arithmetic stress task, respectively and in terms of microbe-brain-gut interactions.

DETAILED DESCRIPTION:
The aim of this study is to determine if and how the "Probiotic Product" affects functional brain responses in healthy subjects during an emotional- and arithmetic stress task, respectively and in terms of microbe-brain-gut interactions.

In this randomized double-blind placebo-controlled study, n=22 healthy subjects will receive the following interventions in a crossover fashion, separated by a 4-week wash-out period: 1) Probiotic Formula, 2) placebo. After baseline assessments, study participants will start with a 4-week intervention with the study product or the placebo, followed by a 4-week wash-out period and a subsequent 4-week intervention period (placebo or study product, respectively). fMRI (functional magnetic resonance imaging) scanning during two validated stress tasks will be performed after each of the intervention periods (week 4 and week 12). At the same time points and in addition on the days before the 1st and 2nd intervention (baseline 1 and 2), saliva, blood and faecal samples will be collected. Questionnaire data will be collected and psychological tests and instruments will be performed. For one week at baseline and during the intervention periods (last week), subjects will wear actigraphs to record their physical activity and help assess sleep quality. At baseline, subjects will undergo a carbon dioxide (CO2) challenge test as well as a food diary to record dietary habits.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Age: 18-65 years, males/females.
2. Signed informed consent -

Exclusion Criteria:

1. Concurrent or recent treatment with drugs affecting intestinal function or mood, e.g., antidepressants (< 12 weeks) or antibiotics (< 12 weeks).
2. Concurrent or recent (< 4 weeks) use of nutritional supplements or herb products affecting intestinal function or mood (e.g. aloe vera, St. John´s Wort, fibers, prebiotics and probiotics).
3. Diagnosis of major psychiatric or somatic disease. 4) Abuse of alcohol or drugs. 5) Recent (< 4 weeks) intake of proton pump inhibitors, proton pump inhibitors, PPIs (e.g., omeprazole).

6) Asthma. 7) Cardiovascular diseases. 8) Epilepsy. 9) Renal failure. 10) Cerebral bleeding or history of cerebral bleeding. 11) Allergic to latex. 12) Pregnancy (assessed by urine test) or breastfeeding. 13) Claustrophobia. 14) Smoking or using tobacco including snuff. 15) Inability to maintain exercise routine and dietary pattern during the study.

16) Consumption of more than 6 cups of coffee/caffeine-containing beverages per day.

17) Professional athlete. 18) Dominant left-hand. 19) Medical implant (e.g., pacemaker). 20) Aneurysm clips in the head. 21) Shunts in the head. 22) Grenade-splinter or metal-splinter in the body (e.g., eyes). 23) Metal or electrodes in the body (e.g., temp-catheter, aorta stent, cochlea implant).

24) Comprehensive tooth-implants or prothesis. 25) Operated in the head. 26) Operated in the heart. 27) Swallowed a video-capsule. 28) Non-corrected astigmatism. 29) Regular intake of systemic corticosteroids and anti-inflammatory medication (including NSAIDs) during the last three months.

30) Visual defect without possibility to use lenses during MRI scanning. 31) Known allergy to milk or soy. 32) Any other reason the investigator feels the subject is not suitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Change in brain response to validated emotional challenge task (EAT) during functional brain imaging | Comparing week 4 and 12

SECONDARY OUTCOMES:
Change in brain response to a cognitive challenge task (MIST) during functional brain imaging | Comparing week 4 and 12

OTHER OUTCOMES:
Change in physical activity assessed by an actigraphy watch (actiwatch) | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Actigraph data regarding physical activity
Change in sleep quality assessed by an actigraphy watch (actiwatch) | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Actigraph data regarding sleep quality
Change in daily stress levels assessed by an actigraphy watch (actiwatch) | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Actigraph data regarding daily stress levels
Autonomous Nervous System (ANS) Activity, Biopac | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  ANS activity is measures during stressful tasks.
Stroop test | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  The Stroop test is performed for stress induction
HADS (Hospital Anxiety and Depression Scale) | Measured weekly, week 1-12
  Hospital Anxiety and Depression Scale, min score 0, max score 3, total score max 42, subscale anxiety max 21, subscale depression max 21
STAI (State and Trait Anxiety Inventory for Adults) | Measured weekly, week 1-12
  State and Trait Anxiety Inventory for Adults
PSS (Perceived Stress Scale) | Measured weekly, week 1-12
  Perceived Stress Scale, min score 0, max score 40
Euro-QoL | Measured weekly, week 1-12
  Euro Qol- Health-related Quality of Life 5Q-5D-5L, min score 0, max score 20, subscale 0-100
Karolinska Sleep Diary (KSD) | Measured daily, week 1-4 and 8-12
  KSD measures sleep quality in the morning
Karolinska Diary of Workload (KDW) | Measured daily, week 1-4 and 8-12
  KDW measures workload daily in the evening
Cortisol levels during fMRI tasks (Saliva) | Comparing week 4 and 12
  Saliva samples are collected during fMRI to assess cortisol levels
Cortisol awakening rhythm (saliva) | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Saliva samples are collected at home (3 days á 5 samples) to assess cortisol levels
Faecal samples | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Faecal samples will be analyzed for quantitative and qualitative microbial composition by 16S rRNA-based next generation sequencing (NGS)
Change in inflammatory markers | Comparing the change in week 0 compared to 4, and 8 compared to 12 (before and in the end of the two intervention periods)
  Blood samples will be collected after each intervention period to assess inflammatory markers using Enzyme-Linked Immunosorbent Assays (ELISA)s

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, Prof, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Campus USÖ, Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rode J, Edebol Carlman HMT, Konig J, Repsilber D, Hutchinson AN, Thunberg P, Andersson P, Persson J, Kiselev A, Lathrop Stern L, Salomon B, Mohammed AA, Labus JS, Brummer RJ. Probiotic Mixture Containing Lactobacillus helveticus, Bifidobacterium longum and Lactiplantibacillus plantarum Affects Brain Responses Toward an Emotional Task in Healthy Subjects: A Randomized Clinical Trial. Front Nutr. 2022 Apr 29;9:827182. doi: 10.3389/fnut.2022.827182. eCollection 2022. PMID 35571902